CLINICAL TRIAL: NCT03110419
Title: Effects of a Multicomponent Training on Postural Control and Cardiovascular and Musculoskeletal Systems in Pre-frail Elderly
Brief Title: Effects of a Multicomponent Training in Pre-frail Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Anielle C M Takahashi, PhD, Adjunt Professor, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAPESI-02
Record Dates: First submitted 2016-08-18; First posted 2017-04-12 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pre-frail Elderly
Keywords: Elderly; Frailty; Multicomponent training; Physical exercise; Functional capacity; Complexity; Physical Therapy
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The training group will perform a Physical Exercise as multicomponent training.
  Interventions: Other: Physical Exercise
- Control (No Intervention): The control group will only be evaluated, without any intervention.

INTERVENTIONS:
Other: Physical Exercise — The intervention program will follow the recommendations of the American College of Sports Medicine (ACSM, 2009), including aerobic, muscle strength, flexibility and balance exercise. The duration of the intervention will be 16 weeks with sessions 60 min performed in three alternate days.
  Other Names: Multicomponent exercise training
  Arms: Intervention

SUMMARY:
This study aim to evaluate the effects of 16 weeks of multicomponent training on postural control, cardiovascular and musculoskeletal systems in pre-frail elderly through nonlinear and linear measurements.

DETAILED DESCRIPTION:
Frailty syndrome is described as a clinical state of vulnerability to stress resulting from the decline of resilience and physiological reserves associated with aging. It is also characterized by a reduction of the interaction between systems and that would be reflected by a loss of physiological complexity. Physical exercise, especially the multi-component, is pointed out as a key element in the intervention of frail elderly individuals. However, it is still unclear whether the improvement in functional capacity observed with this type of training would be related to changes in the physiological complexity of these elderly individuals. The aim of this study is to evaluate the effect of multi-component training on the dynamics of the cardiovascular, motor, neuromuscular and physical activity levels of pre-frail elderly. Thirty-six pre-frail elderly individuals will be divided into intervention (IG, n = 18) and control (CG, n = 18) groups at three different moments (pre-intervention, post-intervention, 16 weeks, and follow-up of detraining of 6 Weeks). The complexity will be evaluated by calculating the entropy of the biological signals: a) heart rate, blood pressure (in supine and orthostatic conditions), b) oscillations of the pressure center (in open, closed eyes, after standing in a chair And under dual-task cognitive condition), c) torque oscillations of the knee extensor muscle group.

ELIGIBILITY:
Inclusion Criteria:

* >= 65 years old;
* conventional ECG without alterations in rest;
* medical release for physical exercise;
* understand the instructions and agree to participate.

Exclusion Criteria:

* historical stroke which produces loss of strength and aphasia;
* several impairment of motor skills;
* Parkinson disease;
* Diabetes Mellitus;
* Peripheral Neuropathy;
* Vestibular and visual disorders self-reported in anamnesis;
* Severe cognitive impairment;
* Cardiovascular disorders (atrial fibrillation, malignant ventricular arrhythmia; ventricular beats complexes ectopic, sinus tachycardia or supraventricular, second and third degree of atrioventricular block, use of pacemaker in the resting ECG);
* Unstable angina;
* Myocardial infarction;
* Elderly end stage.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Linear and nonlinear measurements of postural control | Change from baseline sample entropy and approximate entropy at 16 weeks of multicomponent training and after 6 weeks of detraining
  Sample Entropy; Approximate Entropy
Linear and nonlinear measurements of cardiovascular system | Change from baseline heart rate variability and conditional entropy at 16 weeks of multicomponent training and after 6 weeks of detraining
  Heart Rate Variability; Conditional Entropy
Linear and nonlinear measurements of musculoskeletal systems | Change from baseline knee extensor torque complexity at 16 weeks of multicomponent training and after 6 weeks of detraining
  Knee extensor torque complexity
Cognition Measures | Change from baseline addenbrooke's cognitive examination at 16 weeks of multicomponent training and after 6 weeks of detraining
  Addenbrooke's Cognitive Examination

SECONDARY OUTCOMES:
Functional Measures | Change from baseline six-minute walk test at 16 weeks of multicomponent training and after 6 weeks of detraining
  Six-minute Walk Test
Functional Measures | Change from baseline short physical performance battery at 16 weeks of multicomponent training and after 6 weeks of detraining
  Short Physical Performance Battery

CONTACTS AND LOCATIONS:
Overall Officials: Anielle CM Takahashi, PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carnavale BF, da Silva Santos VR, Farche ACS, Rossi PG, Fiogbe E, de Souza Buto MS, de Vassimon-Barroso V, de Medeiros Takahashi AC. Effects of a multicomponent training and detraining on frailty status, physical activity level, sedentary behavior patterns and physical performance of pre-frail older adults: a randomized controlled trial. Eur Geriatr Med. 2024 Dec;15(6):1701-1712. doi: 10.1007/s41999-024-01052-4. Epub 2024 Sep 11. PMID 39259383